CLINICAL TRIAL: NCT05184153
Title: Medullary Colonic Carcinoma
Acronym: MEDCCR
Status: Completed | Type: Observational
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Other Study IDs: 87RI20_0072 (MEDCCR)
Record Dates: First submitted 2021-10-28; First posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-09

CONDITIONS: Medullary Carcinoma of Colon; Prognostic Factors; Survival Analysis
Keywords: Medullary Carcinoma of Colon; prognostic factors; survival analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Retrospective cohort of 10 cases of colonic adenocarcinoma of medullary type, operated between 2000 and 2020 at the University Hospital of Limoges. Collection of relevant data for this rare entity. Subgroup analysis in search of prognostic factors. Comparison of the data from our cohort with those from the literature.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is the third most common cancer in the world after breast and prostate cancer (1). It is also the second most common cause of cancer death in France (2). Most CRCs are adenocarcinomas. However, there is a distinct subtype of adenocarcinoma of relatively recent recognition, called medullary carcinomas (MC). Its recent recognition as a distinct entity (3) has made it difficult to study the epidemiologic characteristics of this cancer, with little population-based data. The largest cohort studied in the literature is from a US sample of 74 patients seen between 1973 and 2006 (4). The main objective of this French retrospective study is to highlight some common features in this group of patients with medullary colorectal cancers, thus improving our knowledge of this cancer subtype and in particular its prognosis.

Medullary colorectal cancer is a type of cancer with a prognosis of its own, probably different from the most common histological entity, colorectal adenocarcinoma.

This is a retrospective study a cohort of 10 cases of colonic adenocarcinoma of medullary type, operated between 2000 and 2020 at the University Hospital of Limoges. A collection of relevant data was realised for the subgroup analysis in search of prognostic factors for this rare entity as well as a comparison of the data from this cohort with those from the literature.

ELIGIBILITY:
Inclusion Criteria:

* Pathological diagnosis of colorectal adenocarcinoma of medullary type between 2000 and 2020

Exclusion Criteria:

* Absence of anatomopathological confirmation on the surgical specimen

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with an anatomopathological diagnosis of colorectal adenocarcinoma of medullary type managed at the chu de Limoges between 2000 and 2020
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2020-03-03 (Actual); Primary Completion 2020-12-19 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Survival | Through study completion in April 2021
  Number of days between diagnosis and death

SECONDARY OUTCOMES:
Progression | Through study completion in April 2021
  Number of days between first surgery and appearance of metastases

CONTACTS AND LOCATIONS:
Overall Officials: Niki CHRISTOU, Dr, Principal Investigator — 0 33 5 55 05 67 30
Locations (1):
- Service de Chirurgie Digestive et Endocrinienne du CHU de Limoges, Limoges, France